CLINICAL TRIAL: NCT00177814
Title: Piperacillin as a Part of Antibiotic Streamlining in the Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB # 0508074
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Gram-negative Bacterial Infections
Keywords: pipercillin; gram negative bacteria infections
MeSH Terms: conditions — Gram-Negative Bacterial Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The proposed endpoints of the study would be: comparative use of piperacillin versus broader spectrum agents (e.g., piperacillin/tazobactam, etc.) [measured as defined daily doses per 1000 patient days]; physician acceptance of piperacillin as part of a streamlining program [measured as successful occurrences of the use of piperacillin as streamlining therapy]; changes in susceptibility patterns of broad spectrum antibiotics [measured as % Gram negative bacilli susceptible to each of the commonly used broad spectrum antibiotics]; and outcome of patients treated with streamlined therapy.

DETAILED DESCRIPTION:
The following variables will be followed: time and location of positive cultures, underlying diseases and severity of illness, recent immunomodulative therapies, physical exam findings, laboratory and radiographical data, antimicrobial usage, microbiological data and resistance patterns, choice of antibiotics once organism is identified, suspected source of infection, bacteriological outcomes, laboratory results, demographic information, medications, clinical outcome, gender, height, weight, ethnicity, and past medical history.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Gram negative infections treated with piperacillin/tazobactam and/or piperacillin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients treated with piperacillin/tazobactam and or piperacillin
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2005-09 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
dead or alive | end of study
  health status

CONTACTS AND LOCATIONS:
Overall Officials: David Paterson, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States